CLINICAL TRIAL: NCT04061824
Title: Open-label, Randomized, Single Center, Paralleled Clinical Study to Evaluate Adherence Improvement Fixed-dose Combination of Olostar Tab. in Patients With Hypertension and Dyslipidemia
Brief Title: Clinical Study to Evaluate Adherence Improvement Fixed-dose Combination of Olostar Tab. in Patients With Hypertension and Dyslipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4-2015-1122
Record Dates: First submitted 2019-07-26; First posted 2019-08-20 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Hypertension; Dyslipidemias
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — olmesartan; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Intervention Model Description: Patients are divided into 2 group, one with fixed-dose combination of 2 drugs, while another with 2 separated drugs.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with fixed-dose combination of 2 drugs (Experimental): Medication for hypertension and dyslipidemia in these group was fixed-dose combination of 2 drugs
  Interventions: Drug: Olostar Tab (olmesartan/rosuvastatin FDC(fixed dose combination))
- Patients with 2 separated drugs (Active Comparator): Medication for hypertension and dyslipidemia in these group was 2 separated drugs for each disease.
  Interventions: Drug: Two separated drugs(ARB(Angiotensin Ⅱ receptor blocker) and statin)

INTERVENTIONS:
Drug: Olostar Tab (olmesartan/rosuvastatin FDC(fixed dose combination)) — In intervention group, patients had a pill of fixed-dose combination of Olmesartan medoxomil and Rosuvastatin, rather taking separated two pills.
  Arms: Patients with fixed-dose combination of 2 drugs
Drug: Two separated drugs(ARB(Angiotensin Ⅱ receptor blocker) and statin) — In control group, patients had two separated pills for hypertension and dyslipidemia. One of ARBs(Valsartan, Olmesartan, Candesartan, Telmisartan, Fimasartan, Losartan and Irbesartan) and one of statins(Rosuvastatin, Atorvastatin, Pitavastatin, Simvastatin, Pravastatin, Fluvastatin and Atorvastatin/Ezetimibe).
  Arms: Patients with 2 separated drugs

SUMMARY:
Hypertension and dyslipidemia are very prevalent diseases in general population, and the prevalence is keep increasing especially on population with advanced age. Both diseases are major risk factor of cardiovascular disease, and many complication could be induced if not managed properly. Also, these diseases need consistent medication for long time, so the compliance to the treatment is an important issue for these diseases.

Treatment effect of olmesartan to hypertension and rosuvastatin to dyslipidemia is already proven in previous studies, and these medication does not have interaction with each other. By using fixed-dose combination of these drugs, the investigators could improve the compliance to medication, and may have better treatment effect.

In this single center, randomized, phase 4 clinical trial, the investigators divided patients into 2 groups, one with fixed-dose combination of 2 drugs, while another with 2 separated drugs. Each patient in this study was evaluated at first visit, and outcomes are evaluated at 26 weeks after the start point of medication. The primary outcome of this study was compliance of prescribe medication, and the secondary outcome was blood pressure (systolic, diastolic), cholesterol, and low density lipoprotein cholesterol.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between 20 to 80 years old
2. Patients with at least one condition below

   * Systolic blood pressure is 140mmHg or higher, or diastolic pressure is 90mmHg or higher, and 2 or more cardiovascular risk factor, and low-density lipoprotein cholesterol is 130mg/dL or higher.
   * Systolic blood pressure is 140mmHg or higher, or diastolic pressure is 90mmHg or higher, and 0 or 1 cardiovascular risk factor, and low-density lipoprotein cholesterol is 160mg/dL or higher.
   * Patients with medication for hypertension, and (a) symptomatic coronary artery disease, stroke, peripheral artery disease regardless of low density lipoprotein cholesterol level, or (b) diabetes mellitus, carotid artery stenosis of 50% or higher, aortic aneurysm with low density lipoprotein cholesterol 100mg/dL or higher, or (c) more than 2 cardiovascular risk factor with low density lipoprotein cholesterol 130mg/dL or higher, or (d) 0 or 1 cardiovascular risk factor with low density lipoprotein cholesterol 160mg/dL or higher
   * Patients with medication for dyslipidemia, and systolic blood pressure is 140mmHg or higher or diastolic blood pressure is 90mmHg or higher
   * Patients with medication for hypertension and dyslipidemia
3. Patients who can understand the provided information, and sign the consent form

Exclusion Criteria:

1. Systolic blood pressure is 180mmHg or higher, or diastolic blood pressure is 100mmHg or higher
2. Patient with endocrinologic or metabolic disorder which could affect serum lipid or lipoprotein

   - Uncontrolled diabetes mellitus (HbA1c result at baseline evaluation is 9% or higher, or fasting glucose is 160mg/dL or higher
3. Severe cardiologic disorder (heart failure with NYHA class 3 or 4, heart attack in 6 months, myocardial infarction, heart surgery, percutaneous coronary intervention, unstable angina) or coronary artery bypass surgery in 3 months
4. Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically significant cardiac arrhythmia judged by the researcher
5. Patient with genetic disease such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
6. Patient with psychotic disease, or drug or alcohol addiction
7. Patient with severe liver cirrhosis, renal failure, or heart failure
8. Patient with systemic infectious disease
9. Patient who had systemic steroid (intravenous, intramuscular, or per oral) within 2 months before screening, or planned to
10. Patient in pregnancy, lactation, or childbearing age without proper contraceptive measure
11. Patient who attended other clinical trial 1 month before screening
12. Patient who seems to be inappropriate to be in clinical trial judged by researcher

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Compliance of prescribed medication - By using the number of prescribed pills and remained pills, the percentage of admitted drugs were calculated | 26 weeks after the start point of medication
  Compliance of prescribed medication is compared between 2 groups at 26 weeks after the start point of medication. By using the number of prescribed pills and remained pills, the percentage of admitted drugs were calculated.

SECONDARY OUTCOMES:
Blood pressure (systolic, diastolic) | 26 weeks after the start point of medication
  Blood pressure(systolic, diastolic) is compared between 2 groups at 26 weeks after the start point of medication
Cholesterol (mg/dL) | 26 weeks after the start point of medication
  Cholesterol(mg/dL) is compared between 2 groups at 26 weeks after the start point of medication
Low density lipoprotein cholesterol (mg/dL) | 26 weeks after the start point of medication
  Low density lipoprotein cholesterol(mg/dL) is compared between 2 groups at 26 weeks after the start point of medication

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital, Yonsei University Health System, 50 Yonsei-ro, Seodaemun-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No